CLINICAL TRIAL: NCT03168113
Title: Skin Barrier in Childhood Atopic Dermatitis With and Without Food Allergy (ADRN-10)
Brief Title: Atopic Dermatitis (AD) and Food Allergy
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Atopic Dermatitis Research Network (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT ADRN-10
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Atopic Dermatitis (AD); Non-atopic Healthy Controls
Keywords: skin barrier function; microbiome; transepidermal water loss (TEWL); epidermal transcriptome; epidermal lipid composition
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, DNA, Skin tape strip samples and any derivatives, Skin swabs and any derivatives, Stool samples and any derivatives
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AD and Peanut Food Allergy: Participants with active Atopic Dermatitis (AD) and food allergy to peanut.* Twenty participants ages 4 to 17 years of age will be enrolled in this group.
  *Peanut skin prick test wheal ≥ 8 mm.
- AD and No Food Allergy: Participants with active Atopic Dermatitis (AD) and no food allergy.* Twenty participants ages 4 to 17 years of age will be enrolled in this group.
  *Negative skin prick test (wheal < 3 mm) to peanut, milk, egg, wheat, soy, shellfish mix, tree nuts, and sesame seed.
- Non-Atopic Health Control: Participants that are non-atopic, healthy controls*. Twenty participants ages 4 to 17 years of age will be enrolled in this group.
  *Negative for Atopic Dermatitis (AD), asthma, or allergic rhinitis; negative for food allergy; and negative by skin prick test to peanut, milk, egg, wheat, soy, shellfish mix, tree nuts, and sesame seed, and negative to environmental allergens - cat, dog, dust mite, cockroach, and local trees/grasses/weeds/molds.

SUMMARY:
This is a prospective, single center, clinical mechanistic pilot clinical research study. Participants will not receive any investigational agent. The investigators will examine whether children with atopic dermatitis (AD) and food allergy have a different skin barrier, microbiome, epidermal transcriptome, and epidermal lipid composition than children with AD and no food allergy and non-atopic (NA) children. Participation involves a single study visit.

DETAILED DESCRIPTION:
Atopic Dermatitis (AD) is a chronic inflammatory skin disorder in which the skin becomes extremely itchy and is susceptible to recurrent skin infections. AD is thought to occur from a combination of immunological, genetic, and environmental factors.

Those with atopic dermatitis (AD) often have food allergy and Staphylococcus aureus (S. aureus) colonization of the skin. There is evidence suggesting that skin barrier dysfunction, measurable as increased transepidermal water loss (TEWL), is a predisposing factor to food sensitization and food allergy from epicutaneous penetration of environmental food allergens. Furthermore, the investigators for this study have identified that AD children with food allergy, especially peanut allergy, are colonized with Staphylococcus aureus. However, only half (50%) of children with AD have food allergy or S. aureus colonization, suggesting there are other factors accounting for food allergy. There have been no previous studies of TEWL or, microbial or molecular profiling of the skin in those with AD prone to food allergy versus AD without food allergy.

ELIGIBILITY:
Inclusion Criteria:

Participants fulfilling all of the following criteria are eligible for enrollment-

-Parent/guardian must be able to understand and provide informed consent and participant provide assent as applicable per Institutional Review Board (IRB) guidelines and regulations;

For Eligibility to One of the Two Active Atopic Dermatitis (AD) Groups:

-Active Atopic Dermatitis (AD) without a history or current manifestations of eczema herpeticum (EH), as diagnosed using the Atopic Dermatitis Registry

Network (ADRN) Standard Diagnostic Criteria and food allergy to peanut. Participant must meet all of the following criteria:

* Self-report or documentation of a positive oral food challenge to peanut or self-report of an allergic reaction to peanut within 2 hours of ingestion
* Peanut skin prick test wheal ≥ 8 mm. OR -Active AD without a history or current manifestations of EH, as diagnosed using ADRN Standard Diagnostic Criteria and no food allergy.

Participant must meet all of the following criteria:

* No personal history or current manifestations of food allergy (based on no self-report of a positive oral food challenge, positive skin test, positive blood test, or allergic reactions).
* Negative skin prick test (wheal < 3 mm) to peanut, milk, egg, wheat, soy, shellfish mix, tree nuts, and sesame seed.

For Non-atopic (NA) Group Eligibility:

Participant must meet all of the following criteria:

* No personal history or current manifestations of AD, asthma, or allergic rhinitis (based on self-report);
* No personal history or current manifestations of food allergy (based on no self- report of a positive oral food challenge, positive skin test, positive blood test, or allergic reactions);
* Negative skin prick test (wheal < 3 mm) to peanut, milk, egg, wheat, soy, shellfish mix, tree nuts, and sesame seed; and
* Negative skin prick test (wheal < 3 mm) to environmental allergens (cat, dog, dust mite, cockroach, and local trees/grasses/weeds/molds).

Exclusion Criteria:

* Inability or unwillingness of a parent/guardian to give written informed consent, or participant to give assent, if applicable, or to comply with study protocol;
* Subjects with skin disease other than AD that might compromise the stratum corneum barrier (e.g., bullous diseases, psoriasis, cutaneous T cell lymphoma [also called Mycosis Fungoides or Sezary syndrome], dermatitis herpetiformis, Hailey- Hailey, or Darier's disease);
* Pregnant or lactating females;
* Known or suspected immunosuppression;
* Severe concomitant illness(es);
* History of serious life-threatening reaction to latex, tape, or adhesives;
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study;
* Use of biologics within 5 half-lives (if known) or 16 weeks of the Screening Visit;
* Use of an investigational drug within 5 half-lives (if known) or 8 weeks of the Screening Visit; or
* Has received immunotherapy within 12 months of the Screening Visit.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children ages 4-17 years, inclusive. Enrollment will include 20 AD children with food allergy to peanut, 20 AD children without a history of food allergy, and up to 20 NA children. The study requires that AD participants with peanut allergy meet the 95% positive predictive value for skin prick test (≥ 8 mm wheal) for peanut allergy. Food allergic AD participants will be allowed to have other food allergies in addition to peanut. A subset of children with AD whose disease is too severe to stop prohibited medications as defined in the protocol will be excluded. NA children will serve as a healthy control group for the AD study participants. Enrollment is to children since AD and food allergies are more prevalent among children, and adult onset AD and/or food allergy is a different phenotype.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
The Transepidermal Water Loss (TEWL) Area Under the Curve | Visit 1 (Day 1)
  TEWL will be assessed on non-lesional skin prior to tape stripping (Basal) and repeated after 5, 10, 15, and 20 tape strips. TEWL is a noninvasive in vivo measurement of water loss across the stratum corneum. Skin tape strip method allows characterization of components of the epidermis, dermis, and immune cells present in the skin. Comparison between groups (e.g., atopic dermatitis [AD] children with food allergy, AD children without food allergy and Non-atopic children) will be evaluated.

SECONDARY OUTCOMES:
Basal Transepidermal Water Loss (TEWL) | Visit 1 (Day 1)
  TEWL is a noninvasive in vivo measurement of water loss across the stratum corneum that is used to characterize skin water barrier function. Basal TEWL =baseline measure. Comparison between groups (e.g., atopic dermatitis [AD] children with food allergy, AD children without food allergy and Non-Atopic children) of basal TEWL on non-lesional and lesional skin will be evaluated.
Transepidermal Water Loss (TEWL) Measured After 20 Tape Strips | Visit 1 (Day 1)
  TEWL will be assessed on non-lesional skin after 20 tape strips. TEWL is a noninvasive in vivo measurement of water loss across the stratum corneum. Skin tape strip method allows characterization of components of the epidermis, dermis, and immune cells present in the skin. Comparison between groups (e.g., atopic dermatitis [AD] children with food allergy, AD children without food allergy and Non-atopic children) will be evaluated.
Lipid Profiles | Visit 1 (Day 1)
  Lipids, which play a role in the skin barrier, will be extracted from the skin tape strips and measured using mass spectrometry methodology. Sampling will involve the upper extremities. Skin tape strip method allows characterization of components of the epidermis, dermis, and immune cells present in the skin. Comparison between groups (e.g., atopic dermatitis [AD] children with food allergy, AD children without food allergy and Non-atopic children) will be evaluated.

OTHER OUTCOMES:
EXPLORATORY: Protein Expression Profiles | Visit 1 (Day 1)
  Differences between groups (e.g., atopic dermatitis [AD] children with food allergy, AD children without food allergy and Non-atopic children) in protein expression (e.g., proteomic profiles) in samples extracted from skin tape strips will be evaluated. Sampling will involve the upper extremities. Skin tape strip method allows characterization of components of the epidermis, dermis, and immune cells present in the skin. The protein expression profiles will be measured by mass spectrometry of skin tape strips.
EXPLORATORY: Gene Expression Profiles | Visit 1 (Day 1)
  Differential expression of gene transcripts between groups (e.g., atopic dermatitis [AD] children with food allergy, AD children without food allergy and Non-atopic children) will be evaluated from skin tape strips. Skin tape strip method allows characterization of components of the epidermis, dermis, and immune cells present in the skin.
EXPLORATORY: Microbial Carriage | Visit 1 (Day 1)
  Microbial carriage as assessed by the presence of microbial sequencing reads. Skin swab samples will include defined non-lesional and lesional areas of the upper and lower extremities. Comparison of the skin microbiome composition between groups (e.g., atopic dermatitis [AD] children with food allergy, AD children without food allergy and Non-atopic children) using metagenomics.
EXPLORATORY:Carriage of Transcriptionally Active Microbial Species | Visit 1 (Day 1)
  A metatranscriptomics approach will allow for evaluation of the transcriptional response of active microbiome members of the skin. Skin swab samples will include defined non-lesional and lesional areas of the upper and lower extremities. The comparison using this methodology is between groups (e.g., atopic dermatitis [AD] children with food allergy, AD children without food allergy and Non-atopic children).
EXPLORATORY: Frequency of Commensal Antimicrobial Coagulase-Negative Staphylococcus (CoNS) | Visit 1 (Day 1)
  Skin surface bacteria will be collected and typed. Skin swab samples will include defined non-lesional and lesional areas of the upper and lower extremities.
  Comparison between groups (e.g., atopic dermatitis [AD] children with food allergy, AD children without food allergy and Non-atopic children) for anti- Staphylococcus aureus (S. aureus) activity of CoNS cultured from skin will be evaluated. This is a functional assessment of antimicrobial activity.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Leung, M.D., Ph.D., Principal Investigator — National Jewish Health: Division of Pediatric Allergy and Clinical Immunology
Locations (1):
- National Jewish Health: Division of Pediatric Allergy and Clinical Immunology, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data in ImmPort [https://immport.niaid.nih.gov/ ], a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts, upon completion of the study.

REFERENCES:
- [Derived] Lyubchenko T, Collins HK, Goleva E, Leung DYM. Skin tape sampling technique identifies proinflammatory cytokines in atopic dermatitis skin. Ann Allergy Asthma Immunol. 2021 Jan;126(1):46-53.e2. doi: 10.1016/j.anai.2020.08.397. Epub 2020 Sep 5. PMID 32896640
- See also: National Institute of Allergy and Infectious Diseases (NIAID) Website — http://www.niaid.nih.gov/